CLINICAL TRIAL: NCT05670613
Title: Does a Clinical Support System for Parenteral Nutrition (PN) Facilitate the Judgement on Choosing the Most Effective Commercial Solution Per Patient (and Modify it, if Necessary)? Is This Solution an Appropriate Alternative to Customized PN for Optimum Nutrition Outcome?
Brief Title: Does a Clinical Support System for Parenteral Nutrition (PN) Facilitate the Judgement on Choosing the Most Effective Commercial Solution Per Patient (and Modify it, if Necessary)?
Acronym: CDSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Responsible Party: Principal Investigator, Panos Papandreou, Head of Parenteral Nutrition unit, PharmD, Iaso Maternity Hospital, Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19042020
Record Dates: First submitted 2022-11-17; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Clinical Decision Support System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dispense Ready to Use PN Solutions (Other): Dispensed to patient commercial solution.
  Interventions: Other: CDSS Canceling
- Dispense the most effective commercial Solution calculated with the use of the CDSS (Other): Dispensed to patient the most effective commercial solution after the CDSS calculations.
  Interventions: Other: CDSS Canceling

INTERVENTIONS:
Other: CDSS Canceling — The use of Clinical Decision Support System in Parenteral Nutrition

SUMMARY:
Standard formulas of PN have been developed and provided to patients. Only few randomized controlled studies compared standardized vs individualized PN. Individually tailored PN, only if standard PN solutions do not meet patient's nutritional needs. ASPEN society recommends the use computerized prescribing. Technology has enabled the incorporation of medical guidelines in CDSSs. New approach: Comparison of patient's calculated nutritional needs with commercial available solutions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalize Patients unable to be fed via gastrointestinal tract.
* Hemodynamically stable patients.
* PN regimen should remain the same for the first 3 days.

Exclusion Criteria:

* Hemodynamically unstable.
* Anticipated need for parenteral nutrition less than 5 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Estimate of Macro and Micro Nutrient Needs for PN. | 0 months - 12 months
  Estimation of macro and micro nutrient needs for PN by CDSS: amino acids, carbohydrates, lipid, electrolytes, energy and fluids.
Estimate the difference between actual PN energy needs (kcal per day) and energy provided in the PN solutions available in the market (kcal per 100ml). | 0 months - 12 months
  Compare Ready to Use PN solutions with patient's actual nutritional energy needs in order to customize PN for optimum nutrition outcome.
Estimate the difference between actual PN needs and nutrient content of Ready to use Solution for PN available in the market. | 0 months - 12 months
  Compare Ready to Use PN solutions on total grams of amino acids with patient's actual nutritional needs on total grams of amino acids in order to optimize patient's PN for better nutritional outcome.
Estimate the difference between actual PN needs and nutrient content of Ready to use Solution for PN available in the market. | 0 months - 12 months
  Compare Ready to Use PN solutions on total grams of fat with patient's actual nutritional needs on total grams of fat in order to optimize patient's PN for better nutritional outcome.
Estimate the difference between actual PN needs and nutrient content of Ready to use Solution for PN available in the market. | 0 months - 12 months
  Compare Ready to Use PN solutions on total grams of carbohydrates with patient's actual nutritional needs on total grams of carbohydrates in order to optimize patient's PN for better nutritional outcome.
Difference of time spent on estimation of PN needs when conducted by hand and CDSS. | 0 months - 12 months
  Compare time spent for a) calculation of nutritional needs, b) prescription and c) transcription by using CDSS or made by hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Iaso General Hospital, Athens, Greece